CLINICAL TRIAL: NCT00189189
Title: Parent Management Training to Prevent Oppositional Defiant and Conduct Disorders in Preschool Children
Brief Title: Prevention of Oppositional Defiant and Conduct Disorders in Preschool Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 03-119; ZonMw: 2620.0001
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2007-10-02 (Estimated); Status verified 2005-07

CONDITIONS: Oppositional Defiant Disorder; Conduct Disorder
Keywords: prevention; oppositional defiant disorder; conduct disorder
MeSH Terms: conditions — Oppositional Defiant Disorder; Conduct Disorder

INTERVENTIONS:
Behavioral: parent management training

SUMMARY:
Oppositional defiant and conduct disorders are the most frequent bases for referral of children and adolescents. These disorders are difficult to treat among school-aged children and adolescents. When they become adults they are likely to manifest depressive disorders, substance abuse or dependence, and criminal behavior. These disorders are also two of the costly childhood disorders. The aim of the study is to assess the preventive effect of parent management training in preschool children at risk for oppositional defiant and conduct disorders because of high aggression scores on a parent questionnaire. It is hypothesized that given the relatively restricted costs of the intervention and the substantial costs of burden associated with these children, the intervention will be cost saving.

DETAILED DESCRIPTION:
Oppositional defiant and conduct disorders are the most frequent bases for referral of children and adolescents. These disorders are difficult to treat among school-aged children and, even more, among adolescents. When they become adults they are likely to manifest depressive disorders, substance abuse or dependence, criminal behavior and social maladjustment. As parents they are likely to pass along antisocial behavior to their offspring. These disorders are also two of the costly childhood disorders. The children and their parents frequently use social and mental health services. The prevention of these disorders in preschool children at risk thus is clearly relevant.

The origins of oppositional defiant and conduct disorders lie in temperamental vulnerabilities of the preschool child in interaction with non-optimal characteristics of the child's environment. Specifically, ineffective parenting plays a key role in the development of the disorders: a predisposing temperament evokes the kinds of coercive, harsh, inconsistent and negative parenting behaviors that transform a difficult temperament into antisocial behavior. These inadequate parenting behaviors are targeted in parent management training.

In the present study, we will assess the preventive effects of the Incredible Years parent program (Webster-Stratton) in preschool children at risk of oppositional defiant and conduct disorders. Besides, we will study the moderating effects of psychophysiological (heart rate, skin conductance) and neuropsychological variables on intervention outcome. We also will study mediation, i.e. whether the positive outcome is caused by favourable changes in the parenting skills. Finally, costs and cost-effectiveness will be studied.

A hundred sixty children aged four and a half years are selected on the basis of high aggression scores on the Child Behavior Checklist. The parents of seventy children participate in a group parent training. Ninety children serve as care as usual controls and are matched on a person to person basis. Assessments are at pretreatment, posttreatment, one year follow-up, and two year follow-up. Outcome measures consist of parent questionnaires (e.g. CBCL, Eyberg), parent interviews (DDI, DISC), teacher questionnaires (e.g. TRF), and observations of parent-child interactions at home (DPICS). Parenting skills are assessed using observations of parent-child interactions (DPICS). Detailed information on the costs of the intervention and on the costs generated by the conduct problems (medical consumption, education) is monitored.

If the Incredible Years program is shown to be effective, we will have a program in the Netherlands to prevent oppositional defiant and conduct disorders from developing in high-risk preschool children. Four to five year old children who according to their parents or teachers are hard to manage and show high aggression scores on the CBCL or TRF can be monitored. If the scores remain high, the parents are invited to participate in the Incredible Years parent program.

ELIGIBILITY:
Inclusion Criteria:

* Aggression score on Child Behavior Checklist (CBCL) of at least 80th percentile
* Age of child: between 4 and 5 years old

Exclusion Criteria:

* Mastery of the Dutch language is sufficient among the parents to participate in the parent management training

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2003-07; Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Composite score consisting of DPICS (behavioral observation) and parent questionnaires (CBCL, Eyberg)
Teacher questionnaire (TRF)

SECONDARY OUTCOMES:
Cost-effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Walter Matthys, M.D., Ph.D., Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Centre Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Webster-Stratton C, Hammond M. Treating children with early-onset conduct problems: a comparison of child and parent training interventions. J Consult Clin Psychol. 1997 Feb;65(1):93-109. doi: 10.1037//0022-006x.65.1.93. PMID 9103739